CLINICAL TRIAL: NCT03728751
Title: Optimal Time for In-situ Dry Needling to Affect the Autonomic Nervous System: A Pilot Study
Brief Title: Optimal Time for In-situ Dry Needling to Affect the Autonomic Nervous System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida Gulf Coast University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FGCU IRB 2018-51
Record Dates: First submitted 2018-10-29; First posted 2018-11-02 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-10

CONDITIONS: Healthy
Keywords: Dry needling; Autonomic nervous system; pupillometry
MeSH Terms: interventions — Dry Needling

STUDY DESIGN:
Intervention Model Description: Single group pre-test post test study design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study group (Experimental): Study group receiving dry needling and pupil diameter will be studied up to 23 minutes after needle placement.
  Interventions: Procedure: Dry needling

INTERVENTIONS:
Procedure: Dry needling — Paravertebral dry needling C7-T4. Total of 8 needles.

SUMMARY:
Assessing for optimal time dry needles need to remain inside the body to have positive effect on the nervous system

DETAILED DESCRIPTION:
The purpose of this study is to determine what most optimal dry needling duration effect on the autonomic nervous system.

Design: The researchers will conduct a pilot study to assess the effect of dry needling on the autonomic nervous system

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-65 years old
2. No pain at all anywhere in the body at the time of testing.
3. No caffeine containing products 3 hours before measurement and no use of over the counter Non-Steroidal Anti-Inflammatory Drug (NSAID) before the testing.

Exclusion Criteria:

1. Red flags identified during the subjects intake. If needling is contraindicated the subjects will be removed from the study and if necessary will be referred to an appropriate health care provider.
2. Use of blood thinners
3. History of surgery and or injury within the past six weeks
4. Evidence of central nervous system involvement, to include hyperreflexia, sensory disturbances in the hand, intrinsic muscle wasting of the hands, unsteadiness during walking, nystagmus, loss of visual acuity, impaired sensation of the face, altered taste, the presence of pathological reflexes (i.e. positive Hoffman's and/or Babinski reflexes), etc.
5. Prior surgery to the neck or thoracic spine
6. Chiropractic, Physical Therapy, Dry needling or Acupuncture treatment for their neck pain in the last 3-months
7. Inability to follow directions and keep the eye open during the measurement phase of this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2018-10-29 (Actual)

PRIMARY OUTCOMES:
Pupil diameter | 1.) 1 minute measure will be taken after accommodation of 2 minutes to the dark environment, 2.) needle placement and an immediate 1 minute second measure, 3.) every 2 minutes a measure of 1 minute to 8 post needle measures (24 minutes) total
  Change in pupil diameter measured with automated pupillometry device from Micromedical.

CONTACTS AND LOCATIONS:
Overall Officials: Rob Sillevis, PhD, Principal Investigator — Faculty
Locations (1):
- Integrated Therapy Practice PC, Hobart, Indiana, United States

IPD SHARING:
Plan to Share IPD: No